CLINICAL TRIAL: NCT04329754
Title: Safety and Efficacy of a Novel Hydrophobic Acrylic IOL - iPure: a Randomised Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vienna Institute for Research in Ocular Surgery (Other)
Responsible Party: Principal Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Head of Ophthalmology Department, principal investigator, Vienna Institute for Research in Ocular Surgery
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Viros_iPure
Record Dates: First submitted 2013-01-25; First posted 2020-04-01 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — Cataract Extraction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- iPure (Other): A new single-piece hydrophobic acrylic IOL (IPure IOL). The study IOL is a one-piece aspheric acrylic hydrophobic glistening-free lens, with a 4.9% water content, a 360 square posterior edge design, and a 5 haptic angulation, providing UV and blue-light filtration.
  Patient were allocated into two groups. The study group received the iPure lens while the control group received Tecnis ZCB00. Randomisation was done with a binomial law, using random.org. The surgeon was masked to IOL allocation until shortly before implantation. Examiners were masked to IOL allocation.
  Interventions: Device: Cataract surgery
- ZCB00 (Other): A standard IOL (ZCB00).The control IOL, is a one-piece hydrophobic acrylic IOL with a biconvex aspheric optic and 360 continuous square posterior optic edge with a UV filter and an offset, stepped haptic design.
  Patient were allocated into two groups. The study group received the iPure lens while the control group received Tecnis ZCB00. Randomisation was done with a binomial law, using random.org. The surgeon was masked to IOL allocation until shortly before implantation. Examiners were masked to IOL allocation.
  Interventions: Device: Cataract surgery

INTERVENTIONS:
Device: Cataract surgery — Cataract surgery with implantation of an intraocular lens (IOL)

SUMMARY:
In this study the rotational stability and performance - with respect to glistening and PCO formation - of a new hydrophobic acrylic IOL (IPure, PhysIOL, Belgium) will be compared to a gold standard IOL (AMO ZCB00) in a randomized controlled fashion. Fifty eyes of 50 patients will be included. 25 patients will receive the iPure and 25 patients will receive the standard IOL. Study hypothesis: The iPure IOL shows better rotational stability compared to the standard IOL. A clinically relevant difference for rotational stability is defined as 2°.

DETAILED DESCRIPTION:
Although there may be no direct benefit to the subjects under study, the investigation will assess the stability which determines the efficacy for future toric optics and the amount of glistening and PCO formation of the IPure and ZCB00 hydrophobic acrylic IOLs.

25 eyes of 25 patients will be recruited for each IOL, that is 50 eyes of 50 patients. The randomization will be done with a binomial law. The IOL have a priori the same IOL constants which eliminates the necessity to know which IOL is going to be implanted at the preoperative time. A clinically relevant difference for rotational stability will be 2°. The reasonable standard deviation of the position of an IOL in the eye is 2.4°. A total of 48 patients is necessary for a probability of 80% to measure a clinically relevant difference concerning the IOL stability.

In the week before surgery, the eye to be operated is examined at the slit-lamp and by indirect fundoscopy and measurement of intraocular pressure (IOP) will be performed routinely. Additionally, routine biometry is performed using the IOLMaster (Zeiss Meditec AG, Jena, Germany) for axial length measurement, K-readings and anterior chamber depth (ACD) measurements.

Randomisation will be performed using online randomisation and patients will be allocated 1:1 either to the study group (iPure group), or to the control group (ZCB00).

A self sealing incision, injection of viscoelastic substance, capsulorhexis, phacoemulsification, irrigation/aspiration of cortical material and injection of viscoelastic substance into the capsular bag are performed in a standardised fashion. The IOL is implanted via injector into the capsular bag. Following the implantation of the IOL, the viscoelastic substance is aspirated thoroughly from the anterior chamber, as well as retro-lentally, to assure complete removal of the OVD.

Any deviation from the standard protocol will be recorded peroperatively. Follow-ups will be performed 1-2 hours, 1 month, 12 months and 24 months after cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age-related cataract
* Age 21 and older
* Visual Acuity > 0.05
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant.

Exclusion Criteria:

* Relevant other ophthalmic diseases such as pseudoexfoliation syndrome, floppy iris syndrome, corneal pathologies
* Previous ocular surgery or trauma.
* Pregnancy (pregnancy test will be taken pre-operatively in women of reproductive age)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2012-04; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Rotational Stability | 2 years
  measured using the Purkinje meter (Murcia University) and retroillumination images (degrees of rotation)

SECONDARY OUTCOMES:
Glistening | 2 years
  subjective measurement (0 to 4, 0 no glistening, 4 sever glistening)
visual acuity | 2 years
  assessed by ETDRS charts at 4m
PCO | 2 years
  scored with AQUA (0 to 10, 0 no PCO, 10 sever PCO) and the number of Nd:YAG capsulotomies
Decentration in mm | 2 years
  measured by Purkinjemeter
Tilt in degrees | 2 years
  measured by Purkinjemeter
Capsulorhexis area | 2 years
  assessed by retroillumination images
Anterior chamber depth | 2 years
  assessed by AC Master (in mm)

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Findl, MD, MBA, Principal Investigator — VIROS, Hanusch Hospital Vienna
Locations (1):
- Vienna Institute for Research in Ocular Surgery (VIROS), Hanusch Hospital Vienna, Vienna, Austria